CLINICAL TRIAL: NCT01452074
Title: Progressive Metabolic Adaptations to Low Intensity Exercise Training and Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeffrey F Horowitz, Associate Professor, Movement Science, School of Kinesiology, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R01 DK077966 - PA; R01DK077966 (NIH)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Insulin Sensitivity; Exercise Training; Weight Loss; Fat Metabolism
MeSH Terms: conditions — Obesity; Insulin Resistance; Weight Loss | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Training with Weight Loss (Other): During the first 12 weeks of the study, subjects will adhere to an exercise training program while maintaining their original body weight. The exercise training program will entail the following: 40min/session, ~50% of their maximal aerobic capacity (approximately 100-110 beats per min), 5-6 days/week
  After the first 12 weeks in the study, subjects will continue with the same exercise program, but then they will be placed on a reduced calorie diet until they lose exactly 10% of their original body weight
  Interventions: Other: Exercise Training; Other: Weight Loss with continued Exercise Training

INTERVENTIONS:
Other: Exercise Training — During the first 12 weeks of the study, subjects will adhere to an exercise training program while maintaining their original body weight. The exercise training program will entail the following: 40min/session, ~50% of their maximal aerobic capacity (approximately 100-110 beats per min), 5-6 days/week
Other: Weight Loss with continued Exercise Training — After the first 12 weeks in the study, subjects will continue with the same exercise program, but then they will be placed on a reduced calorie diet until they lose exactly 10% of their original body weight

SUMMARY:
the investigators first aim is to determine the effect of low intensity exercise (without weight loss) on insulin sensitivity, muscle lipid metabolism, and factors regulating these processes in skeletal muscle after 1 day, 2 wks, 12 wks of training, and again after 3 days without exercise in obese adults. the investigators second aim is to determine the effect of combining low intensity exercise training with 10% weight loss on insulin sensitivity, muscle lipid metabolism, and factors regulating these processes in skeletal muscle.

Although a single 40 minute session of exercise at a low exercise intensity will not improve insulin sensitivity, the investigators anticipate adaptations after two weeks of exercise training (6 session/wk; 12 session total) will improve insulin sensitivity and be accompanied by a reduction in fatty acid intermediates and a reduction in markers for pro-inflammatory activation in muscle. the investigators anticipate changes in insulin sensitivity, fatty acid partitioning, and pro-inflammatory markers the day after the last session of a 12 wk training program (without weight-loss) will be similar to that measured after 2 weeks of training. the investigators anticipate insulin sensitivity, accumulation of fatty acid intermediates, and pro-inflammatory activation will be markedly improved after 10% weight loss when measured the day after exercise. the investigators would expect the improvements in Insulin sensitivity, accumulation of fatty acid intermediates, and markers of inflammatory stress will be significantly attenuated when measured 3 days after the most recent exercise session, but beneficial effects of 10% weight loss on these metabolic endpoints will persist when compared with before weight loss.

ELIGIBILITY:
Inclusion Criteria:

* body mass index [BMI]: 30-45 kg/m2; All women must be pre-menopausal; Non-exerciser (no regularly planned exercise/physical activity)

Exclusion Criteria:

* Hematocrit ≤ 34%; Fasting plasma glucose concentration ≥ 125 mg/dL; Weight instability ≥ ±5 lbs in past month; Taking medications known to affect lipid and/or glucose metabolism; evidence and/or history of cardiovascular or frank metabolic diseases; pregnancy or actively breast feeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-07-18 (Actual); Study Completion 2014-07-18 (Actual)

PRIMARY OUTCOMES:
Insulin Sensitivity | 2-3 hours
  A hyperinsulinemic-euglycemic clamp will be used to assess peripheral insulin sensitivity

SECONDARY OUTCOMES:
Resting Metabolic Rate | 20-30 min
Meal Tolerance Test | 2-3h

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Horowitz, Principal Investigator — University of Michigan
Locations (1):
- Michigan Clincal Research Unit, Ann Arbor, Michigan, United States